CLINICAL TRIAL: NCT02565264
Title: Effect of Plasma Derived Exosomes on Intractable Cutaneous Wound Healing: Prospective Trial
Brief Title: Effect of Plasma Derived Exosomes on Cutaneous Wound Healing
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kumamoto University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2019-09

CONDITIONS: Ulcer
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- plasma-derived exosomes (Experimental): plasma-derived exosomes
  Interventions: Other: plasma-derived exosomes

INTERVENTIONS:
Other: plasma-derived exosomes — Plasma samples from the participants will be filtered through 0.45 μm and 0.20 μm filters. The samples will be filtered through 0.02 μm filter to trap exosomes with the filter. Saline solution will be loaded from the other side of the 0.02 μm filter to obtain exosome rich buffer. The plasma-derived exosomes will be applied to the participants' ulcers daily for 28 days.

SUMMARY:
This study is an open prospective clinical trial. The objective is to evaluate the effect of autologous exosomes rich plasma on cutaneous wound healing. The participants are patients with intractable cutaneous ulcers (e.g. rheumatic disease, peripheral arterial disease, chronic venous insufficiency, decubitus or burns). The participants will be treated autologous exosomes rich plasma every day for 28 days. The cutaneous wound healing will be evaluated by the length, width and depth of the wound.

DETAILED DESCRIPTION:
Exosomes are small vesicles 0.03-0.1 μm in size, which are shed from most cell types into the extracellular space via intracellular endocytosis. They are found abundantly in body fluids such as blood. They consist of lipid bilayer so that their structure is stable. They can be preserved for 2 weeks at 4℃. They contain proteins, lipids and nucleic acids including coding or non-coding RNA. Resent studies have revealed that exosomes have an important role in cell-to-cell communication.

The investigators found that serum exosome levels were significantly decreased in scleroderma patients with vascular involvements such as cutaneous ulcers and/or pitting scars compared to in normal subjects. The investigators also elucidated that serum-derived exosomes accelerated cutaneous wound healing in BALB/c mice. Exosome supplementation to cutaneous ulcers seems to have significant therapeutic value.

The objective of present study is to evaluate the effect of exosomes derived from plasma on intractable cutaneous ulcers (e.g. rheumatic disease, peripheral arterial disease, chronic venous insufficiency, decubitus or burns).

Autologous exosomes are obtained from the participants' own plasma. The duration of study is 28days. The cutaneous wound healing will be evaluated at day1, day2, day7, day14, day 21 day 28.

ELIGIBILITY:
Inclusion Criteria:

Patients with intractable cutaneous ulcers (e.g. rheumatic disease, peripheral arterial disease, chronic venous insufficiency, decubitus or burns)

Exclusion Criteria:

1. Patients who have ulcers with bone involvement.
2. Patients who have ulcers with a history or suspected neoplasia.
3. Patients who are in chemotherapy or radiation therapy on the skin ulcers.
4. Patients with marked immunodeficiency (i.e., patients with severe liver failure, heart failure, hematologic failure or endocrine failure)
5. Patients who have clinical signs of malnutrition or serum albumin <2 mg / dL.
6. Patients who have severe infection.
7. Patients who are pregnant or breastfeeding.
8. Patients who are participating in another study.
9. Patients who are judged inappropriate for this trial by their attending physician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Ulcer size (length, mm) | 28 days
Ulcer size (width, mm) | 28 days
Ulcer size (depth, mm) | 28 days

SECONDARY OUTCOMES:
Pain of cutaneous wounds (Visual Analog Score for pain) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jinnin Masatoshi, MD, PhD, Principal Investigator — Department of Dermatology and Plastic Surgery, Faculty of Life Sciences, Kumamoto University
Locations (1):
- Department of Dermatology and Plastic Surgery, Faculty of Life Sciences, Kumamoto University, Kumamoto, Japan